CLINICAL TRIAL: NCT05764980
Title: Assessment Study of Neurovisual Function in CHARGE Syndrome
Brief Title: Neurovisual Function in CHARGE Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Zampino Giuseppe, Associate Professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 3373
Record Dates: First submitted 2023-03-01; First posted 2023-03-13 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: CHARGE Syndrome
Keywords: CHARGE syndrome; Visual function
MeSH Terms: conditions — CHARGE Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: visual function evaluation — visual function evaluation

SUMMARY:
The rationale of the study is to analyze visual function and correlate them with adaptive functions in patients with CHARGE syndrome in order to identify a pattern of specific indicators to enable better patient care

DETAILED DESCRIPTION:
CHARGE syndrome is a malformative condition characterized by coloboma in about 70-95% of patients. This anatomical abnormality results in severe visual impairment that strongly affects the characterization of the disability profile.

Although the ocular anatomical deficits associated with the syndrome have been extensively described in the literature, coloboma being a major criterion for diagnosis, little is reported about the characteristics of visual function, such as acuity, visual field ocular motility, and other features.

Patients with CHARGE syndrome have multiple sensory deficif often accompanied by intellectual disability, which often makes the classical methods used in ophthalmologic evaluation inapplicable. According to the few studies in the literature, visual acuity in patients with CHARGE syndrome is often severely impaired with mean values below 20/60 (McMain et al 2008; Nishina et al 2012; Russell-Eggitt et al. 1990; Stromland et al. 2005; Tellier et al. 1998) However in opposition to the recurrent pessimistic findings resulting from ophthalmologic assessment in clinical practice, such patients present with good visual and adaptive abilities in daily life.

The rationale of the study is to analyze visual function and correlate them with adaptive functions in patients with CHARGE syndrome in order to identify a pattern of specific indicators to enable better patient care

ELIGIBILITY:
Inclusion Criteria:

Patients with molecularly confirmed CHARGE syndrome.

Exclusion Criteria:

Patients with CHARGE syndrome that has not been molecularly confirmed

Ages: 0 Years to 90 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients of all ages with molecularly confirmed CHARGE sidnrome
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-03-15 (Actual); Primary Completion 2023-03-15 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
To demonstrate the correlation between severity of anatomical impairment and neurovisual ability. | 4 years
  to detect aspects of visual function by studying ocular motility, visual acuity, contrast sensitivity, distance attention, and binocular visual field

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Zampino, medicine, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli Irccs, Roma, Italy